CLINICAL TRIAL: NCT03229473
Title: Validity and Reliability of Balance Screening Tests for Fall Risk Assessment in COPD
Brief Title: Fall Risk Assessment in COPD
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: West Park Healthcare Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 3331
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Disease; COPD
Keywords: Balance; Falls; Screening; COPD
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with chronic obstructive pulmonary disease (COPD) have balance problems and are at risk of falling. New guidelines recommend balance assessment be included in pulmonary rehabilitation (PR) however no specific tests are recommended. Our goal is to determine the best balance test for identifying COPD patients who are at risk of falling. In this study, COPD patients who report balance problems or falling in the last year will participate in a testing session. Balance, balance confidence, lower body strength, exercise tolerance and perceived physical limitations will be assessed. The number of falls over the following year will be recorded using monthly calendars.

DETAILED DESCRIPTION:
COPD is a leading cause of death, disability and hospitalization in Canada. In addition to the primary lung impairment, secondary effects of the disease are well established including impairments in muscle function, mobility and exercise capacity. Individuals with COPD also have marked deficits in balance and an increased risk of falls.

The updated American Thoracic Society/European Respiratory Society Statement on PR recommended expanding the scope of outcome assessment in COPD to include balance however no specific tests are suggested. An examination of brief balance measures feasible for fall risk screening has not been conducted. Such information will inform clinicians as to those most likely to benefit from targeted intervention. This study aims to determine the optimal balance measure for identifying patients with COPD who are high risk for falling.

The specific objectives of the study are to: 1) Investigate the construct validity (convergent and known-groups) and reliability (inter-rater and test-retest) of three short balance screening measures in people with COPD; 2) Investigate the predictive validity of the balance screening tests for falls; and 3) Identify cut-off scores for identifying fallers with COPD on the balance screening tool with the strongest psychometric properties.

One hundred and twenty individuals with COPD will be recruited from two sites. Upon enrolment, participants will undergo a physical assessment session measuring balance, functional lower body strength and exercise tolerance. Participants will also complete questionnaires of balance confidence, perceived physical function limitations, fall risk, dyspnea, global cognitive impairment and executive function. Participants will then be followed for 12 months to measure incidence of falls.

To assess inter-rater reliability of the primary measures, two raters will simultaneously administer the balance tests with a subset of the first 32 subjects to agree to participate in this study. This subset will also be asked to return for repeat testing two-three days after the baseline assessment to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD according to GOLD guidelines
* history of one or more falls in the previous year or a self-reported problem with balance/fear of falling
* ability to provide written informed consent

Exclusion Criteria:

* inability to communicate because of language skills (e.g. aphasia, non-English speaking)
* inability to follow instructions due to dementia or severe cognitive impairment
* evidence of a condition that severely limits mobility (e.g Parkinson's disease, cerebrovascular accident)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals greater than 60 years of age diagnosed with COPD who have had one or more falls in the last year or who self-report problems with their balance or fear of falling.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Brief-Balance Evaluation Systems Test (Brief-BESTest) | Upon enrolment, sub-group will repeat 2-3 days later.
  Measure of balance. The Brief-BESTest is a shortened 6-item version of the 36-item full BESTest
Timed Up and Go (TUG) | Upon enrolment, sub-group will repeat 2-3 days later.
  Measure of balance and functional mobility in older adults. Includes a dual-task condition.
Single-leg Stance Test (SLS) | Upon enrolment, sub-group will repeat 2-3 days later.
  Measure of balance.
Incidence of Falls | baseline, 12 months
  Falls during the previous year will be measured at baseline and then prospectively for 12 months using monthly fall diary calendars.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Upon enrolment
  Measure of balance.
Activities-specific Balance Confidence Scale (ABC Scale) | Upon enrolment
  Measure of balance confidence.
30-second Repeated Chair Stand Test | Upon enrolment
  Measure of functional lower body strength.
Six-Minute Walk Test (6MWT) | Upon enrolment
  Measure of exercise tolerance.
Self-reported function (PF-10) | Upon enrolment
  Physical function sub-scale of the Medical Outcomes Study 36-item Short-form Health Survey
Fried's Frailty Phenotype | Upon enrolment
  Measure of frailty including the following criteria: weight loss, exhaustion, physical activity, walk speed and grip strength in community-dwelling older adults.
Mini-Mental State Exam | Upon enrolment
  Measure of five areas of cognitive function: orientation, registration, attention and calculation, recall, and language.
Trail Making Test | Upon enrolment
  Measure of cognitive executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Marla Beauchamp, PhD, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - North Hamilton Community Health Centre, Hamilton, Ontario
  - Firestone Institute for Respiratory Health, Hamilton, Ontario
  - West Park Healthcare Centre, Toronto, Ontario

REFERENCES:
- [Derived] Nguyen KT, Ellerton C, Wald J, Raghavan N, Macedo LG, Brooks D, Goldstein R, Beauchamp MK. Validation of a clinical prediction model for falls in community-dwelling older adults with COPD: A preliminary analysis. Chron Respir Dis. 2025 Jan-Dec;22:14799731251321494. doi: 10.1177/14799731251321494. PMID 39957244